CLINICAL TRIAL: NCT04736186
Title: Prevention and Treatment of Pyrrolitinib-associated Diarrhea: a Prospective, Multicenter, Open-label Clinical Study
Brief Title: Prevention and Treatment of Pyrrolitinib-associated Diarrhea
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YWBC-002
Record Dates: First submitted 2020-09-22; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2020-05

CONDITIONS: Breast Cancer
Keywords: Diarrhea; Non-secondary prevention; Secondary prevention; pyrrolitinib
MeSH Terms: conditions — Breast Neoplasms; Diarrhea | interventions — Loperamide

STUDY DESIGN:
Intervention Model Description: Non-secondary prevention: Explore the recovery time of oral loperamide 4mg T.I.D. for pyrrolitinib induced diarrhea of 1-2 degrees.
  Secondary prevention: To explore the incidence of grade 3 and above diarrhea during c1D1-C1D22 in patients with oral loperamide 4 mg, T.I.D. (D1-7) →4 mg, B.I.D. (D8-21).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Loperamide (Experimental): Loperamide 4 mg, T.I.D. (D1-7) →4 mg, B.I.D. (D8-21)
  Interventions: Drug: Loperamide
- Loperamide and gold bifid (Experimental): Loperamide 4 mg, T.I.D. (D1-7) →4 mg, B.I.D. (D8-21) + gold bifid2g T.I.D.
  Interventions: Drug: Loperamide; Drug: Loperamide and golden bifid
- Loperamide and Montmorillonite SAN (Experimental): Loperamide 4 mg, T.I.D. (D1-7) →4 mg, B.I.D. (D8-21) + Montmorillonite SAN 3 g, T.I.D.
  Interventions: Drug: Loperamide; Drug: Loperamide and montmorillonite powder
- Non-intervention (No Intervention): Do not intervene and stop diarrhea as needed

INTERVENTIONS:
Drug: Loperamide — Loperamide 4 mg， t.i.d.(d 1-7);4 mg, b.i.d.(d 8-21)
  Arms: Loperamide; Loperamide and Montmorillonite SAN; Loperamide and gold bifid
Drug: Loperamide and golden bifid — Patients with secondary prevention will be randomly assigned to B：Loperamide 4 mg， t.i.d.(d 1-7);4 mg, b.i.d.(d 8-21)+golden bifid 2 g t.i.d.
  Arms: Loperamide and gold bifid
Drug: Loperamide and montmorillonite powder — Patients with secondary prevention will be randomly assigned to D：Loperamide 4 mg， t.i.d.(d 1-7);4 mg, b.i.d.(d 8-21)+montmorillonite powder 3 g t.i.d.
  Arms: Loperamide and Montmorillonite SAN

SUMMARY:
In this study, patients taking pyrrolitinib alone or combined with pyrrolitinib were recruited (170 cases of secondary prevention and 300 cases of non-secondary prevention).

Non-secondary prevention: Explore the recovery time of oral loperamide 4mg T.I.D. for pyrrolitinib induced diarrhea of 1-2 degrees.

Secondary prevention: To explore the incidence of grade 3 and above diarrhea during c1D1-C1D22 in patients with oral loperamide 4 mg, T.I.D. (D1-7) →4 mg, B.I.D. (D8-21).

DETAILED DESCRIPTION:
The study can only be formally carried out with the written approval of the ethics committee. Investigators regularly submit annual research reports to the ethics committee. Investigators will inform the ethics committee in writing when the study is discontinued and / or completed.

All patients were required to sign informed consent before entering the group. All updated versions of informed consent and written information will be provided to the subjects during the participant's participation.

In the experimental design stage, the statistical principle was used to make reasonable and effective arrangements for the relevant factors. Employ statistical experts to calculate the sample size and data statistics, and participate in the design process. Data collection and follow-up were conducted by specially assigned personnel, professional doctors were assigned to conduct data review regularly, and special data management personnel were provided. They will ensure the authenticity, reliability and security of data throughout the process.

ELIGIBILITY:
Inclusion Criteria:

1. One of the following two situations:

   A) Plan to take pyrrolitinib for ≥21 days; B) Third-degree diarrhea or second-degree diarrhea with complications after taking pyrrolitinib at present, plan to take pyrrolitinib for ≥21 days;
2. Age ≥18 years;
3. ECOG PS 0-2;
4. Life expectancy ≥6 months;
5. Participate in this study voluntarily, sign informed consent, have good compliance and are willing to cooperate with the follow-up.

Exclusion Criteria:

1. May be allergic to pyrrolitinib or excipients;
2. There are many factors affecting the absorption of oral drugs, such as inability to swallow, nausea and vomiting;
3. Patients with biliary obstruction;
4. Participate in other diarrhea-related clinical trials;
5. Pregnant and lactating women, fertile women who tested positive in the baseline pregnancy test, or women of childbearing age who were unwilling to use effective contraception during the whole trial period;
6. Concomitant diseases (including but not limited to severe hypertension beyond the control of drugs, severe diabetes, etc.) that, according to the judgment of the researcher, seriously endanger the safety of the patient or affect the completion of the study; The investigator concluded that the patient was not eligible for any of the other conditions in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2020-05-16 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
time from the first day of treatment until diarrhea returns to level 0 or baseline during the first day of treatment to the 22nd day of treatment | From the first day of treatment to the 22nd day of treatment(about 21 days)
  Non-secondary prevention
The proportion of 3/4 degree diarrhea in group A From the first day of treatment to the 22nd day of treatment | From the first day of treatment to the 22nd day of treatment(about 21 days)
  Secondary prevention

SECONDARY OUTCOMES:
Loperamide combined program, diarrhea recovery to level 0 or baseline time | From the first day of treatment to the 22nd day of treatment(about 21 days)
  Non-secondary prevention
3/4 degree incidence of diarrhea | From the first day of treatment to the 22nd day of treatment(about 21 days)
  Non-secondary prevention
The accumulated time of diarrhea during the follow-up period | From the first day of treatment to the 22nd day of treatment(about 21 days)
  Non-secondary prevention
Time of first occurrence of diarrhea | From the first day of treatment to the 22nd day of treatment(about 21 days)
  Non-secondary prevention
The incidence rate of all degrees of diarrhea during the follow-up period | From the first day of treatment to the 22nd day of treatment(about 21 days)
  Non-secondary prevention
The incidence of constipation of degree 2 or above during the follow-up period | From the first day of treatment to the 22nd day of treatment(about 21 days)
  Non-secondary prevention
Other AE/SAE during the follow-up period | From the first day of treatment to the 22nd day of treatment(about 21 days)
  Non-secondary prevention
The proportion of cases with 3/4 degree diarrhea | From the first day of treatment to the 22nd day of treatment(about 21 days)
  secondary prevention
The proportion of incidences of 3/4 degree diarrhea during follow-up | From the first day of treatment to the 22nd day of treatment(about 21 days)
  secondary prevention
The incidence rate of all degrees of diarrhea during the follow-up period | From the first day of treatment to the 22nd day of treatment(about 21 days)
  secondary prevention
The incidence of constipation of degree 2 or above during the follow-up period | From the first day of treatment to the 22nd day of treatment(about 21 days)
  secondary prevention
The time of the first diarrhea attack during the follow-up period | From the first day of treatment to the 22nd day of treatment(about 21 days)
  secondary prevention
The cumulative duration of diarrhea during the follow-up period | From the first day of treatment to the 22nd day of treatment(about 21 days)
  secondary prevention
Proportion of subjects with delayed or reduced doses of pyrrolitinib due to diarrhea | From the first day of treatment to the 22nd day of treatment(about 21 days)
  secondary prevention
Other AE/SAE during the follow-up period | From the first day of treatment to the 22nd day of treatment(about 21 days)
  secondary prevention

OTHER OUTCOMES:
Risk factor analysis for diarrhea（The baseline information, demographic data, past treatment history, treatment plan and diet habits of patients with diarrhea were summarized, and the risk factors of diarrhea were summarized） | From the first day of treatment to the 22nd day of treatment(about 21 days)
  exploratory，descriptive results
Analysis of intestinal flora（During the experiment, the feces were collected three times for microbiological examination, and the results of microbiological examination were summarized and analyzed to understand the types of microbiota） | From the first day of treatment to the 22nd day of treatment(about 21 days)
  exploratory，descriptive results
Efficacy of pyrrolitinib (According to the curative effect evaluation standard of solid tumor version 1.1, the imaging curative effect of tumor was evaluated） | From the first day of treatment to the 22nd day of treatment(about 21 days)
  exploratory，descriptive results

CONTACTS AND LOCATIONS:
Locations (1):
- TianJin Medical University Cancer Institute and Hospital, Tianjin, China